CLINICAL TRIAL: NCT00534807
Title: Effect of Rifampin on the Pharmacokinetics of Intravenous (IV) Vinflunine in Subjects With Advanced Cancer
Brief Title: A Study of the Interaction of Rifampin and Vinflunine in Subjects With Advanced Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA183-033
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2007-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — vinflunine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vinflunine
Drug: Rifampin

SUMMARY:
The purpose of this study is to test how vinflunine interacts with rifampin in the human body

ELIGIBILITY:
Inclusion Criteria:

* Cancer unresponsive to previous treatment
* Consent for genetic samples

Exclusion Criteria:

* Cancer of the blood
* Spread of cancer to the brain
* Moderate or severe nerve damage
* Low white blood cell counts and platelet counts
* Inadequate liver or kidney function
* Prior treatment with vinflunine
* Use of certain medications that might interfere with the metabolism of vinflunine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
The Primary Outcome Measure of the effect of rifampin on the pharmacokinetics (PK) of intravenous (IV) vinflunine will be determined from the PK measurements | taken during Cycle 2 of study treatment, at approximately 4 weeks after the start of study treatment

SECONDARY OUTCOMES:
The Secondary Outcome Measures of the safety and tolerability of vinflunine when administered alone and with rifampin | determined after 2 complete 21-day Cycles of study treatment, at approximately 6 weeks after the start of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Detroit, Michigan, United States